CLINICAL TRIAL: NCT07309315
Title: Inactivated Bacteroides Fragilis for Prevention of Chemotherapy-Induced Diarrhea
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Hospital of Southern Medical University (Other)
Responsible Party: Principal Investigator, Hongwei Zhou, Hospital Director, Shenzhen Hospital of Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SK10-IIT
Record Dates: First submitted 2025-12-12; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Chemotherapy-induced Diarrhea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1 (Experimental): Trial Group of Patients with Advanced Colorectal Cancer
  Interventions: Drug: Inactivated Bacteroides fragilis
- Arm 2 (Placebo Comparator): Control Group of Patients with Advanced Colorectal Cancer
  Interventions: Drug: Placebo
- Arm 3 (Experimental): Trial Group of Patients with Breast Cancer
  Interventions: Drug: Inactivated Bacteroides fragilis
- Arm 4 (Placebo Comparator): Control Group of Patients with Breast Cancer
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Inactivated Bacteroides fragilis — Live Biotherapeutic Products
  Other Names: SK10
  Arms: Arm 1; Arm 3
Drug: Placebo — Placebo
  Arms: Arm 2; Arm 4

SUMMARY:
The incidence of chemotherapy-induced diarrhea (CID) is closely related to the types of anticancer drugs. Combination chemotherapy regimens such as fluorouracil derivatives and irinotecan, as well as tyrosine kinase inhibitors like neratinib, are associated with a high severity and incidence of diarrhea. These All antineoplastic agents can induce intestinal epithelial cell apoptosis, damage the intestinal mucosa, subsequently reduce the absorption surface area, and thereby lead to diarrhea. Recent literature has indicated that Bacteroides fragilis may be a candidate drug for the treatment and prevention of CID. This study intends to conduct a randomized controlled trial to determine the efficacy and mechanism of action of inactivated Bacteroides fragilis (SK10) in the prevention of chemotherapy-induced diarrhea (CID).

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form, be able to comply with the protocol and have the capacity to complete relevant procedures.
2. Aged ≥ 18 years old (based on the date of signing the ICF), regardless of gender.
3. Patients with malignant tumors confirmed by pathology or cytology.
4. Patients scheduled to receive the following first-line treatments at the standard dose specified in the protocol:

   * Cohort 1: Patients with advanced colorectal cancer receiving the FOLFIRI regimen (irinotecan + fluorouracil + leucovorin);
   * Cohort 2: Patients with breast cancer receiving neratinib treatment.
5. ECOG performance status score of 0-1 at the start of the study.
6. Expected survival time ≥ 12 weeks.
7. Subjects of childbearing potential (including males and females) agree to adopt effective contraceptive measures approved by the investigators (e.g., intrauterine device, contraceptive pills or condoms) during the trial and within 3 months after the trial ends. Female subjects of childbearing potential must have a negative result in serum human chorionic gonadotropin (hCG) test.

Exclusion Criteria:

1. History of altered bowel habits or abnormal stool characteristics prior to screening; or use of laxatives within 7 days prior to randomization; or use of antidiarrheal agents within 48 hours prior to randomization.
2. Complicated with diseases causing diarrhea, including but not limited to inflammatory bowel disease (e.g., ulcerative colitis and Crohn's disease), suspected or confirmed infectious diarrhea, irritable bowel syndrome, celiac disease, etc.
3. Receipt of any chemotherapeutic agents, cetuximab or PD-1 antibodies other than the chemotherapy/treatment regimen specified in the protocol during the trial.
4. Previous or concurrent abdominopelvic radiotherapy during the trial period.
5. Medical history of chronic use of laxatives (≥ 30 non-consecutive days).
6. Need for antibiotic treatment during the trial or long-term use of antibiotics prior to randomization.
7. Patients with stomas (temporary stomas should be closed for at least 6 months prior to randomization).
8. Presence of unhealed surgical wounds, ulcers or fractures.
9. Known history of human immunodeficiency virus (HIV) infection (positive HIV antibody test).
10. History of allergy or suspected allergy to antidiarrheal drugs (e.g., loperamide and its components).
11. Suspected or confirmed history of alcohol or drug abuse.
12. Pregnant or lactating women.
13. Concurrent participation in other clinical trials.
14. Other conditions deemed inappropriate for study participation by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Overall Incidence of Diarrhea | 4 weeks
  Proportion of Patients with Any Grade of Diarrhea assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Incidence of Grade ≥2 Diarrhea | 4 weeks
  Proportion of Patients with Grade 2 or Higher Diarrhea assessed by CTCAE v5.0
Incidence of Grade ≥3 Diarrhea | 4 weeks
  Proportion of Patients with Grade 2 or Higher Diarrhea assessed by CTCAE v5.0
Days of Diarrhea | 4 weeks
  Mean Days of Diarrhea per Treatment Cycle
Frequency of Diarrhea | 4 weeks
  Mean Frequency of Stool Type 6 or 7 per Treatment Cycle
Percentage and Days of Patients Receiving Antidiarrheal Treatment | 4 weeks
  Percentage of patients treated with antidiarrheal drugs (loperamide, diphenoxylate, octreotide, montmorillonite), defined as the proportion of patients with at least one dose of antidiarrheal drugs relative to the total number of cases; days of antidiarrheal treatment, defined as the mean days of antidiarrheal drug administration per treatment cycle.
Proportion of Patients Who Received Medical Treatment for Diarrhea | 4 weeks
  Proportion of patients who sought medical attention due to diarrhea and received intravenous fluid replacement or anti-infective treatment from investigators.
Proportion of Patients Who Had Chemotherapy/Treatment Dose Reduction, Delay or Discontinuation Due to Diarrhea | 4 weeks
  Proportion of patients with chemotherapy/treatment dose reduction, delay or discontinuation as judged by investigators due to diarrhea.
Relative Dose Intensity of Chemotherapy/Treatment | 4 weeks
  Ratio of delivered dose intensity (mg/m² or mg) to planned dose intensity (mg/m² or mg)
Incidence of Other Gastrointestinal Symptoms | 4 weeks
  Proportion of patients with at least one episode of any grade of gastrointestinal symptoms (constipation, abdominal distension, abdominal pain, hematochezia, nausea, vomiting) assessed by CTCAE v5.0.
Change in Quality of Life Score of Cancer Patients Compared with Baseline | 4 weeks
  Defined as the change in the QLQ-C30 quality of life scale score of cancer patients after study intervention compared with the baseline.
Incidence of Adverse Event (AE) | 4 weeks
  Proportion of participants with adverse events as assessed by CTCAE v5.0
Incidence of Serious Adverse Event (SAE) | 4 weeks
  Proportion of participants with Serious Adverse Event (SAE) as assessed by GCP 2020

OTHER OUTCOMES:
Change in Levels of Blood Inflammatory Cytokines Compared with Baseline | 4 weeks
  Blood inflammatory cytokines Including but not limited to TNF-α, IL-6, IL-1β, IL-4, IL-10, IL-11, etc. Change in Levels of Blood Inflammatory Cytokines Compared with Baseline defined as the change in the levels of blood inflammatory cytokines of cancer patients after study intervention compared with the baseline.
Change in Composition and Diversity of Fecal Flora Structure, and Change in Fecal Metabolomics | 4 weeks
  Change in Composition and Diversity of Fecal Flora Structure defined as the change in the composition and diversity of fecal flora structure of cancer patients after study intervention compared with the baseline.
  Change in Fecal Metabolomics defined as the change in the fecal metabolomics of cancer patients after study intervention compared with the baseline.

IPD SHARING:
Plan to Share IPD: No